CLINICAL TRIAL: NCT00038311
Title: Safety and Efficacy of (PN-152,243)/PN-196,444 in the Prevention of Thrombocytopenia Administered to Patients With High-Risk Sarcoma Receiving Intensive Chemotherapy (Adriamycin and Ifosfamide (AI))
Brief Title: Safety and Efficacy of (PN-152,243)/PN-196,444 in the Prevention of Thrombocytopenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 444-ONC-0003-020
Record Dates: First submitted 2002-05-30; First posted 2002-05-31 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma

INTERVENTIONS:
Drug: PN-152,243)/PN-196,444

SUMMARY:
Intensive chemotherapy is associated with significant thrombocytopenia, often requiring platelet transfusion to maintain platelet counts. This investigational drug has demonstrated the ability to increase platelet counts. This study will test the safety and efficacy of an investigational drug in the prevention of thrombocytopenia in patients with high-risk sarcoma receiving AI (Adriamycin/Ifosfamide) chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be newly diagnosed with moderate or high-grade sarcoma and be receiving AI (Adriamycin/Ifosfamide) chemotherapy

Exclusion Criteria:

* Patients must not have active bleeding (exclusions do apply) or history of platelet disorder

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2000-09; Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness of intravenous rhTPO versus placebo in reducing the cumulative proportion of patients who experience severe chemotherapy induced thrombocytopenia.

SECONDARY OUTCOMES:
Identify the effect of rhTPO on the number of platelet transfusions.
Evaluate the severity and duration of thrombocytopenia and neutropenia associated with rhTPO prophylaxis.
Quantify the effect of rhTPO on the occurrence of any bleeding events associated with thrombocytopenia.
Assess the likelihood that patients were to have adequate hematological recovery to allow on-time chemotherapy administration in the subsequent cycles.
Assess the safety of multiple IV doses of rhTPO.
Determine the occurrence and clinical implications of any anti-TPO antibodies.
Assess the antitumor activity of AI chemotherapy.
Evaluate the impact of rhTPO prophylaxis on health economics/cost effectiveness.
Evaluate the impact of rhTPO prophylaxis on patient quality of life.
Determine serum concentrations of TPO in the context of rhTPO and chemotherapy administration

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (6):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Park Ridge, Illinois
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Radnor, Pennsylvania
  - Pfizer Investigational Site, Houston, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=444-ONC-0003-020&StudyName=Safety+and+Efficacy+of+%28PN%2D152%2C243%29%2FPN%2D196%2C444+in+the+Prevention+of+Thrombocytopenia